CLINICAL TRIAL: NCT01372072
Title: A Pilot Study to Investigate the Physiological and Clinical Effects of Heated Humidification During Non-Invasive Ventilation
Brief Title: A Study to Investigate the Effects of Heated Humidification During Non-Invasive Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RJ1 11/N141
Record Dates: First submitted 2011-06-09; First posted 2011-06-13 (Estimated); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Chronic Obstructive Pulmonary Disease; Chronic Respiratory Hypercapnic Failure; Neuromuscular Disease; Obesity Hypoventilation Syndrome
Keywords: chronic respiratory hypercapnic failure
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Neuromuscular Diseases; Obesity Hypoventilation Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Humidification (Active Comparator): Patients in this arm of the trial will receive humidification with the non-invasive ventilation.
  Interventions: Device: non-invasive ventilation heated humidification (Fisher-Paykel MR810 and MR850 humidifiers)
- NIV without humidifivation (No Intervention): As per usual practice patients in this arm will not have humidification with their NIV

INTERVENTIONS:
Device: non-invasive ventilation heated humidification (Fisher-Paykel MR810 and MR850 humidifiers) — Heated humidification (Fisher-Paykel MR810 and MR850 humidifiers)
  Arms: Humidification

SUMMARY:
Noninvasive ventilation (NIV) is a form of ventilation delivered by a mask and is an important mode of treatment in patients with both acute and chronic respiratory (breathing) failure. Humidification is widely accepted as an essential part of the ventilation strategy in patients receiving invasive ventilation (i.e. via a tube inserted into the mouth), but its role during NIV use is not proven. Consequently, there is a variation in practice with regard to humidification during NIV. Humidification is important in maintaining upper and lower airway mucosal function and patients requiring NIV often report symptoms, such as throat dryness, due to a lack of airway humidity. Success of NIV in the acute setting is dependent on many factors including, patient tolerance of NIV during the acute phase. In patients with chronic obstructive airways disease (COPD), poor tolerance results in NIV failure, which necessitates endotracheal intubation or treatment failure. Furthermore, invasive ventilation increases the risk of a hospital acquired pneumonia, which is associated with a worse outcome. In the long term setting of NIV use, again patients frequently report symptoms due to drying of the airways and adherence to NIV can be highly variable. Adherence in these patients is important in improving both quality and length of life. Humidification devices may be technically effective, but clinicians have concerns regarding potential negative effects of these devices. There is a requirement to evaluate the use of humidification in both the acute and long term use of NIV, particular, in terms of patient ventilator interaction, which will impact on comfort and adherence to NIV. This will effect the overall effectiveness of ventilation. The investigators propose a randomised controlled trial to investigate the effects of a humidification system during noninvasive ventilation.

ELIGIBILITY:
Inclusion Criteria:

* hypercapnic respiratory failure
* age > 18
* requiring non-invasive ventilation

Exclusion Criteria:

* psychiatric illness
* pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2014-09-30 (Actual); Study Completion 2014-09-30 (Actual)

PRIMARY OUTCOMES:
Adherence to NIV | up to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Swapna Mandal, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- St Thomas' Hospital, London, United Kingdom

REFERENCES:
- [Derived] Mandal S, Ramsay M, Suh ES, Harding R, Thompson A, Douiri A, Moxham J, Murphy PB, Hart N. External heated humidification during non-invasive ventilation set up: results from a pilot cross-over clinical trial. Eur Respir J. 2020 May 21;55(5):1901126. doi: 10.1183/13993003.01126-2019. Print 2020 May. No abstract available. PMID 32366486